CLINICAL TRIAL: NCT07092150
Title: Long-term Effectiveness and Implementation of the Meals, Education, and Gardens for In-School Adolescents (MEGA) Program - MEGA 2.0
Brief Title: Long-term Effectiveness and Implementation of the Meals, Education, and Gardens for In-School Adolescents Program
Acronym: MEGA 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: George Mason University (Other); Africa Academy for Public Health (Other); University of Dodoma (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB25-0043
Record Dates: First submitted 2025-07-12; First posted 2025-07-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Anemia; Nutritional Status
Keywords: Randomized controlled trial; Schools; Adolescent nutrition; Tanzania
MeSH Terms: conditions — Anemia | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: The study will have two arms - intervention and control. Four schools will be assigned to the intervention arm, and two schools will be assigned to the control arm. The five components of the proposed intervention package are 1) school feeding, 2) school garden, 3) nutrition education, 4) community workshops, and 5) weekly iron and folic acid (IFA) supplementation and annual deworming. Adolescents in control schools will not receive any of these interventions but will be provided with standard of care practices at secondary schools in Dodoma. In addition, teachers in control schools will receive a hard copy of educational materials on nutrition, agriculture, and WASH to enhance their lesson plans and the community workshop manual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): School meals, gardens, education, iron and folic acid supplementation, and workshops for women.
  Interventions: Other: School meals; Other: School gardens; Dietary Supplement: IFA and Deworming; Behavioral: Nutrition education; Behavioral: Women's workshops
- Control (No Intervention): Standard of care

INTERVENTIONS:
Other: School meals — Daily mid-day meals sourced locally and supplemented by school gardens.
  Arms: Intervention
Other: School gardens — A school vegetable garden to grow green leafy vegetables on school grounds.
  Arms: Intervention
Dietary Supplement: IFA and Deworming — Weekly iron and folic acid supplements and annual deworming.
  Arms: Intervention
Behavioral: Nutrition education — Nutrition education, led by trained teachers, that will cover health, agriculture, and WASH topics.
  Arms: Intervention
Behavioral: Women's workshops — Community workshops that will engage mothers or female guardians in gardening, nutrition, and entrepreneurship, offering support and training for small businesses and homestead gardens.
  Arms: Intervention

SUMMARY:
The overall objective of the proposed study is to determine the longer-term effectiveness and implementation of an updated school-based nutrition intervention package for reducing adolescent malnutrition. Aim 1 of the study is to determine the longer-term effectiveness of an updated intervention package on reducing adolescent malnutrition using a cluster randomized controlled trial in Dodoma, Tanzania. Four intervention schools and two control schools will be included. The intervention schools will receive an intervention package that includes school feeding, nutrition education, school vegetable garden, community workshops, and weekly iron and folic acid supplementation and annual deworming. The control schools will not receive any intervention. The intervention package will be implemented over one year. In each school, 125 adolescents aged between 14 and 17 and 125 mothers/female guardians will be enrolled. The primary outcomes will be moderate to severe anemia in adolescents and underweight in adolescents. The secondary outcomes will include anemia (any severity) and overweight/obesity in adolescents, diet quality in adolescents and mothers/female guardians, household food insecurity, and women's empowerment for mothers/female guardians. A baseline and an end-line evaluation of the outcomes will be implemented. Aim 2 of the study will be to assess the implementation of the updated intervention package by collecting quantitative and qualitative data from adolescents, mothers/female guardians, teachers, smallholder farmers, agricultural extension workers, school administrators, and governmental stakeholders. Using a convergent mixed methods approach, quantitative data (via questionnaires) and qualitative data (via semi-structured interviews and focus group discussions) will be analyzed to evaluate the implementation of the intervention package and identify its implementation barriers and facilitators.

DETAILED DESCRIPTION:
This study will be a cluster-randomized controlled study and will use a mixed-methods approach to evaluate the longer-term effectiveness and implementation of an updated school-based intervention package on adolescent nutritional status in six public secondary schools in Chamwino District, Dodoma, Tanzania. Specifically:

* Aim 1 of the study is to determine the longer-term effectiveness of the updated school-based intervention package on reducing adolescent malnutrition.
* Aim 2 of the study is to assess the implementation of the updated school-based intervention package.

Study Design

This is a two-arm study comparing an intervention group to a control group. Four schools will be assigned to the intervention arm, and two schools will be assigned to the control arm. The study duration is one academic year. Baseline and endline data collection will occur at the beginning and end of the academic year, respectively. Implementation and sustainability data will be collected towards the end of the intervention period.

Intervention Arm (MEGA 2.0 Package)

The MEGA 2.0 intervention is a unified package delivered to adolescents in intervention schools, comprising five integrated components:

* School Feeding: Daily midday meals provided to all adolescents in intervention schools, meeting 60-75% of their daily energy and nutritional requirements. Meals will consist of traditional Tanzanian staples, green leafy vegetables, and will integrate local produce from farm-to-school partnerships and school gardens. School meal committees involving parents, teachers, and administrators will be established to enhance sustainability and community buy-in, with opportunities for mothers to be employed as cooks.
* School Gardens: Establishment of a vegetable garden in each intervention school. Adolescents will participate in gardening activities under the supervision of a trained focal teacher. Agricultural extension workers will provide technical support.
* Nutrition Education: Weekly sessions for adolescents led by focal teachers, covering health and nutrition, agriculture and school gardening, health benefits of vegetables, physical activity and body size, and WASH (Water, Sanitation, and Hygiene).
* Community Workshops: Bi-weekly workshops for mothers and female guardians, conducted by agricultural extension workers. Workshops will utilize school gardens as "model farms" and cover nutrition, agriculture, WASH, and entrepreneurship skills. Participants will receive seeds and gardening supplies as feasible for homestead gardens and guidance on local market entry and microfinancing schemes.
* Weekly Iron and Folic Acid (IFA) Supplementation and Annual Deworming: Weekly IFA supplements will be administered to adolescents by focal teachers during nutrition education sessions. Annual deworming with mebendazole (500 mg) will also be provided.

Control Arm

Adolescents in control schools will not receive any study interventions. They will continue with standard of care practices at secondary schools in Dodoma. Currently, standard of care in Tanzania does not include school meals or government-run school feeding programs in secondary schools. Teachers in control schools will receive a hard copy of educational materials on nutrition, agriculture, and WASH to enhance their lesson plans and a community workshop manual, to use at their discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent Quantitative Survey:

   1. Student enrolled in Form 1 or 2 in a participating school
   2. Between the ages of 14-17
   3. Parent or guardian provides consent for the adolescent
   4. Adolescent provides assent
   5. Fluent in Swahili
2. Adolescent Qualitative Focus Group Discussion (FGD):

   1. Student enrolled in Form 1 or 2 in a participating school
   2. Between the ages of 14-17
   3. Identified by their teacher as a suitable candidate for the focus group
   4. Parent or guardian provides consent for the adolescent
   5. Adolescent provides assent
   6. Fluent in Swahili
3. Mother Quantitative Survey and Qualitative FGD:

   1. Mother or female guardian of participating adolescent
   2. Provides informed consent
   3. Fluent in Swahili
4. Focal Teacher Qualitative Semi-Structured Interview (SSI):

   1. Teacher facilitating the meal, garden, education, and supplementation interventions
   2. Provides informed consent
   3. Fluent in Swahili
5. Smallholder Farmer Qualitative SSI:

   1. Farmers involved in the provision of local produce for school feeding
   2. Provides informed consent
   3. Fluent in Swahili or English
6. Agricultural Extension Worker Qualitative SSI:

   1. Extension workers involved in school garden and community workshops
   2. Provides informed consent
   3. Fluent in Swahili
7. School Administrator Qualitative SSI:

   1. School administrators involved in the intervention
   2. Provides informed consent
   3. Fluent in Swahili

Exclusion Criteria:

Those who do not meet the above listed inclusion criteria.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Selection of adolescents will not be based on gender. However, for parents and guardians, only mothers and female guardians will be invited to participate.
Enrollment: 1500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
1. Moderate to severe anemia in adolescents | Baseline and endline (approximately 12 months after baseline)
  Hemoglobin concentration < 110 g/L in girls and boys
Underweight in adolescents | Baseline and endline (approximately 12 months after baseline)
  BMI-for-age z-score < -2 by WHO growth reference

SECONDARY OUTCOMES:
Anemia (any severity) in adolescents | Baseline and endline (approximately 12 months after baseline)
  Hemoglobin concentration < 120 g/L in girls and < 130 g/L in boys
Overweight or obesity in adolescents | Baseline and endline (approximately 12 months after baseline)
  BMI-for-age z-score ≥ 1 by WHO growth reference
Diet quality of adolescents | Baseline and endline (approximately 12 months after baseline)
  Diet quality as defined by the Global Diet Quality Score; a higher score indicates a better diet quality
Diet quality of mothers | Baseline and endline (approximately 12 months after baseline)
  Poor diet quality as defined by the Global Diet Quality Score; a higher score indicates a better diet quality
Household food insecurity | Baseline and endline (approximately 12 months after baseline)
  Defined by Household Food Insecurity Access Scale; a higher score indicates more severe food insecurity
Women's empowerment in mothers | Baseline and endline (approximately 12 months after baseline)
  Defined by the Abbreviated Version of the Women's Empowerment in Agriculture Index (A-WEAI); a higher score indicates greater empowerment

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, MPH, MS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Dongqing Wang, PhD, MPH, Principal Investigator — George Mason University
Locations (1):
- University of Dodoma, Dodoma, Tanzania

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Wang D, Katalambula LK, Modest AR, Ismail A, Malero A, Bray D, Cinq-Mars H, Tinkasimile A, Sando MM, Vuai S, Fawzi WW. Meals, Education, and Gardens for In-School Adolescents: A Cluster Randomized Trial of an Adolescent Nutrition Intervention Package in Tanzania. J Adolesc Health. 2024 Jul;75(1):115-126. doi: 10.1016/j.jadohealth.2024.02.032. Epub 2024 Apr 8. PMID 38597842